CLINICAL TRIAL: NCT00516048
Title: An Exploratory Study of the Effect of Treatment Interruption on Safety of Exenatide in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8O-MC-GWBO
Record Dates: First submitted 2007-08-10; First posted 2007-08-14 (Estimated); Results first posted 2009-06-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: exenatide; Byetta; antibodies; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide:Treatment-Emergent Antibody Negative (Experimental): This arm will receive 5mcg exenatide for 4 weeks, followed by 10mcg exenatide for 20 weeks.
  Interventions: Drug: exenatide
- Exenatide:Treatment-Emergent Antibody Positive (Experimental): This arm will receive 5mcg exenatide for 4 weeks, followed by 10mcg exenatide for 20 weeks.
  Interventions: Drug: exenatide

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, 5mcg or 10mcg, twice a day
  Other Names: Byetta; AC2993; LY2148568

SUMMARY:
The primary purpose of this study is to assess the anti-exenatide-antibody response to exenatide re-exposure as measured by anti-exenatide antibodies and incidence of treatment-emergent allergy and hypersensitivity reactions following a period of treatment interruption, in patients previously exposed to exenatide.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes.
* Have been exposed to exenatide for at least 3 months in previous Amylin/Lilly Studies H8O-MC-GWAO, H8O-MC-GWAP, H8O-MC-GWAT, or H8O-MC-GWBA.
* Have interrupted exenatide treatment for a period of at least 2 months.
* HbA1c of ≤10.5%.

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Have previously completed or withdrawn from this study.
* Have taken marketed exenatide (Byetta) during the interim period between studies GWAO, GWAP, GWAT, or GWBA and the current study.
* Used drugs for weight loss (for example, Xenical® [orlistat], Meridia® [sibutramine], Acutrim® [phenylpropanolamine], Accomplia® [rimonabant], or similar over-the-counter medications) within 3 months of screening.
* Are currently treated with any of the following excluded medications: Drugs that directly affect gastrointestinal motility, including, but not limited to: Reglan® (metoclopramide), Propulsid® (cisapride), and chronic macrolide antibiotics.
* Use insulin with daily dosage exceeding 1 U/kg.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (13):
- Research Site, Keswick, South Australia, Australia
- Canada (3):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, London, Ontario
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Gyula
  - Research Site, Zalaegerszeg
- Italy (3):
  - Research Site, Milan
  - Research Site, Perugia
  - Research Site, Rome
- South Korea (3):
  - Research Site, Seonnam City
  - Research Site, Seoul
  - Research Site, Suwon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following a period of treatment interruption of at least 2 months, patients for this study were recruited from among patients who were previously exposed to exenatide for at least 3 months in Amylin/Lilly studies GWAO, GWAP, GWAT, and GWBA.
Groups:
- Exenatide:Treatment-Emergent Antibody Negative: 5mcg exenatide for 4 weeks, followed by 10mcg exenatide for 20 weeks. Assessed as negative for antibodies to exenatide throughout the study.
- Exenatide: Treatment-Emergent Antibody Positive: 5mcg exenatide for 4 weeks, followed by 10mcg exenatide for 20 weeks. Assessed as positive for antibodies to exenatide at any point in the study.
- Enrolled But Withdrew Before Receiving Treatment: No exenatide treatment administered and no post-baseline (post-Week 0) assessment of antibody status was conducted.
Period: Overall Study
Arm/Group | Exenatide:Treatment-Emergent Antibody Negative | Exenatide: Treatment-Emergent Antibody Positive | Enrolled But Withdrew Before Receiving Treatment
Started | 15 | 42 | 1
Completed | 15 | 40 | 0
Not Completed | 0 | 2 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Subject Decision | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Negative Baseline (Week 0) Antibody Status: Patients assessed as negative for antibodies to exenatide at baseline (Week 0).
- Positive Baseline (Week 0) Antibody Status: Patients assessed as positive for antibodies to exenatide at baseline (Week 0).
- Total: Total of all reporting groups
Arm/Group | Negative Baseline (Week 0) Antibody Status | Positive Baseline (Week 0) Antibody Status | Total
Number analyzed (Participants) | 50 | 8 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 8 | 39
  >=65 years | 19 | 0 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.65 (8.95) | 49.88 (9.84) | 59.17 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 5 | 25
  Male | 30 | 3 | 33

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Antibody Status (Maximum Titer Level Experienced)
Description: Patients who experienced specified treatment-emergent antibody status at any point during the study (grouped by maximum titer level experienced)
Time Frame: 24 weeks
Population: Intent to Treat
Measure: Number; unit: Participants
Arm/Group | Exenatide:Treatment-Emergent Antibody Negative | Exenatide: Treatment-Emergent Antibody Positive | Enrolled But Withdrew Before Receiving Treatment
Number analyzed (Participants) | 15 | 42 | 1
Participants
  Antibody negative | 15 | 0 | 0
  Low titer antibodies | 0 | 25 | 0
  Higher titer antibodies | 0 | 17 | 0

2. Secondary Outcome: Change in Hemoglobin A1c (HbA1c) From Baseline to Endpoint
Description: Change in HbA1c from baseline (Week 0) to endpoint (Week 24) by treatment-emergent antibody status
Time Frame: 24 weeks
Population: Intent to Treat; Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Exenatide:Treatment-Emergent Antibody Negative | Exenatide: Treatment-Emergent Antibody Positive | Enrolled But Withdrew Before Receiving Treatment
Number analyzed (Participants) | 15 | 42 | 1
percent
  Baseline HbA1c (Week 0) | 8.13 (0.66) | 8.05 (1.00) | 0 (0)
  Change in HbA1c at endpoint (Week 24) | -1.03 (0.74) | -0.30 (0.94) | 0 (0)

3. Primary Outcome: Incidence of Potentially Immune-related Treatment-emergent Adverse Events
Description: Number of patients experiencing a potentially immune-related treatment-emergent adverse event at any point during the study
Time Frame: 24 weeks
Population: Intent to Treat
Measure: Number; unit: participants
Arm/Group | Exenatide:Treatment-Emergent Antibody Negative | Exenatide: Treatment-Emergent Antibody Positive | Enrolled But Withdrew Before Receiving Treatment
Number analyzed (Participants) | 15 | 42 | 1
participants
  Arthralgia | 1 | 0 | 0
  Spinal osteoarthritis | 1 | 0 | 0
  Injection site pruritis | 0 | 2 | 0
  Injection site rash | 0 | 1 | 0
  Rash | 0 | 1 | 0
  Eye allergy | 0 | 1 | 0

ADVERSE EVENTS:
Arm/Group | Exenatide:Treatment-Emergent Antibody Negative | Exenatide: Treatment-Emergent Antibody Positive | Enrolled But Withdrew Before Receiving Treatment
Serious Adverse Events (participants affected / at risk) | 0 | 1 | 1
Other Adverse Events (participants affected / at risk) | 7 | 11 | 0
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Exenatide:Treatment-Emergent Antibody Negative | Exenatide: Treatment-Emergent Antibody Positive | Enrolled But Withdrew Before Receiving Treatment
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/15 | 1/42 | 0/1
Sudden death (General disorders) | 0/15 | 0/42 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Exenatide:Treatment-Emergent Antibody Negative | Exenatide: Treatment-Emergent Antibody Positive | Enrolled But Withdrew Before Receiving Treatment
Nasopharyngitis (Infections and infestations) | 1/15 | 2/42 | 0/1
Influenza (Infections and infestations) | 0/15 | 2/42 | 0/1
Injection site pruritis (General disorders) | 0/15 | 2/42 | 0/1
Toothache (Gastrointestinal disorders) | 0/15 | 2/42 | 0/1
Viral infection (Infections and infestations) | 0/15 | 2/42 | 0/1
Diarrhoea (Gastrointestinal disorders) | 1/15 | 1/42 | 0/1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/15 | 0/42 | 0/1
Gastrooesphageal reflux disease (Gastrointestinal disorders) | 1/15 | 0/42 | 0/1
Hyperglycaemia (Metabolism and nutrition disorders) | 1/15 | 0/42 | 0/1
Otitis externa (Infections and infestations) | 1/15 | 0/42 | 0/1
Otitis media (Infections and infestations) | 1/15 | 0/42 | 0/1
Periodontitis (Gastrointestinal disorders) | 1/15 | 0/42 | 0/1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/15 | 0/42 | 0/1
Vomiting (Gastrointestinal disorders) | 1/15 | 0/42 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days